CLINICAL TRIAL: NCT00004685
Title: Randomized Study of Albuterol in Patients With Facioscapulohumeral Muscular Dystrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/13285; OSURF-96H0022; OSURF-FDR001293
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 1999-03

CONDITIONS: Muscular Dystrophy, Facioscapulohumeral
Keywords: genetic diseases and dysmorphic syndromes; muscular dystrophy; neurologic and psychiatric disorders; rare disease
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral; Genetic Diseases, Inborn; Muscular Dystrophies; Neurologic Manifestations; Mental Disorders; Rare Diseases | interventions — Albuterol

INTERVENTIONS:
Drug: albuterol

SUMMARY:
OBJECTIVES: I. Determine whether albuterol increases strength in patients with facioscapulohumeral dystrophy as measured by quantitative voluntary isometric contraction testing.

II. Determine whether albuterol increases muscle mass in this patient population as determined by 24 hour urinary creatinine excretion and dual energy x-ray absorptiometry (DEXA).

III. Examine the long term safety of albuterol in this patient population.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double blind, placebo controlled study. Patients are randomized into one of three treatment groups. The first group receives placebo. The second group receives low dose albuterol orally every 12 hours. The third group receives high dose albuterol orally every 12 hours. Treatment continues for 52 weeks unless unacceptable side effects occur.

All patients return for follow up assessments at weeks 4, 12, 24, and 52.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Facioscapulohumeral dystrophy Weakness of the facial muscles, including frontalis, orbicularis oculi, or orbicularis oris Weakness of scapular stabilizers or foot dorsiflexors Weakness of grade 2 or worse in the arm using the upper extremity grading scale No other neuromuscular diseases that may mimic the clinical presentation of facioscapulohumeral dystrophy: Ptosis or ophthalmoparesis (other than congenital strabismus) Elbow contractures Strictly unilateral weakness Dermatomyositis-like skin rash Symmetric distal sensory loss Muscle biopsy findings of mitochondrial myopathy, chronic denervation, dermatomyositis, inclusion body myositis, or congenital myopathy Electromyographic (EMG) findings of myotonia, fasciculations, or neurogenic motor unit potentials --Prior/Concurrent Therapy-- Endocrine therapy: No prior long term use of oral corticosteroids for more than 1 year At least 3 months since prior use of corticosteroids No concurrent use of immunosuppressive agents Surgery: No concurrent surgeries Other: No concurrent use of sympathomimetic agents, antidepressants, or beta receptor blockers --Patient Characteristics-- Age: 18 to 80 Performance status: Ambulatory Cardiovascular: No cardiovascular disease, including hypertension and coronary artery disease Other: Not pregnant or nursing No concurrent uncontrolled medical or psychological condition

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 1998-01; Study Completion 2000-09

CONTACTS AND LOCATIONS:
Overall Officials: John T. Kissel, Study Chair — Ohio State University